CLINICAL TRIAL: NCT00468741
Title: Component and Couple Analysis of Cancer Communications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2003-193; 1P50CA09817-01A1 (Other Grant/Funding Number: National Cancer Institute); CC04318 (Other: University of Wisconsin, Madison); 2003-193 (Other: Institutional Review Board); A534253 (Other: UW Madison); SMPH/MEDICINE/MEDICINE (Other: UW Madison)
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Internet; Computer; Support; Information; Education; Control Group: Usual care and Internet access; CHESS Information Services only; CHESS Social Support & Information Services; CHESS Information, Social Support & Skills Services
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention): subjects receive internet access and computer
- 2 (Experimental): CHESS informational services only
  Interventions: Behavioral: CHESS
- 3 (Experimental): CHESS social support and informational services
  Interventions: Behavioral: CHESS
- 4 (Experimental): Full CHESS
  Interventions: Behavioral: CHESS (Comprehensive Health Enhancement Support System)

INTERVENTIONS:
Behavioral: CHESS (Comprehensive Health Enhancement Support System) — Full CHESS for subject use
  Arms: 4
Behavioral: CHESS — informational services of CHESS available to subject
  Arms: 2
Behavioral: CHESS — CHESS informational services and social support available to subject
  Arms: 3

SUMMARY:
Component and Couple Analysis of Cancer Communication

CHESS, the Comprehensive Health Enhancement Support System is an innovative technology that provides information, social support and skills training to women with breast cancer. Previous CHESS clinical trials found improved patient outcomes but little is known about what services in CHESS produce those results. This study will examine whether breast cancer patient outcomes change when conceptually distinct CHESS services (information, social support, and skills training) are systematically added to a patients treatment resources.

Primary Aims:

* Determine the relative efficacies of different types of cancer communication treatments when they are presented alone or in combination
* Determine routes or processes via which these elements work
* Determine for whom the different treatment types work best.

ELIGIBILITY:
Inclusion Criteria:

Eligibility for this protocol is as follows:

* All subjects must be within 2 months of their primary breast cancer diagnosis,
* All subjects must be at least 18 years of age,
* All subjects must be able to read and write English at the 6th-grade level
* Not homeless

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2003-09; Primary Completion 2008-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patient Quality of Life | monthly

SECONDARY OUTCOMES:
Emotional Well-being | monthly
Self Efficacy | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - M. D. Anderson, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/